CLINICAL TRIAL: NCT05126329
Title: An Open-label Pharmacokinetic and Tolerability Study of Amcenestrant Given as a Single Dose in Female Participants With Mild and Moderate Hepatic Impairment, and in Matched Participants With Normal Hepatic Function
Brief Title: Pharmacokinetics of Amcenestrant in Female Hepatic Impaired Participants as Compared to Participants With Normal Hepatic Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP16301; U1111-1244-1929 (Registry Identifier: ICTRP); 2021-001784-24 (EudraCT Number)
Record Dates: First submitted 2021-11-03; First posted 2021-11-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Function Abnormal
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with mild hepatic impairment (Experimental): Amcenestrant 200 mg single dose on Day 1 in fed condition
  Interventions: Drug: amcenestrant
- Participants with moderate hepatic impairment (Experimental): Amcenestrant 200 mg single dose on Day 1 in fed condition
  Interventions: Drug: amcenestrant
- Participants with normal hepatic function (Experimental): Amcenestrant 200 mg single dose on Day 1 in fed condition
  Interventions: Drug: amcenestrant

INTERVENTIONS:
Drug: amcenestrant — tablet for oral use

SUMMARY:
This is a Phase 1, parallel, open-label, 3-arm study to investigate the pharmacokinetic (PK) parameters of amcenestrant in female participants aged 40 to 75 years with mild and moderate hepatic impairment, and in matched participants with normal hepatic function.

DETAILED DESCRIPTION:
The total study duration from screening period is approximately 41 days.

ELIGIBILITY:
Inclusion Criteria:

For participants with hepatic impairment:

* Participant must be 40 to 75 years of age, inclusive.
* Female participants who are postmenopausal or are post-bilateral surgical oophorectomy not linked to a history of cancer. Menopause is defined as being amenorrheic for at least 12 months without an alternative medical cause, with plasma FSH level >30 IU/L or age ≥60 years.
* Stable chronic liver disease assessed by medical history, physical examination, laboratory values
* Body weight within the range 50 kg (40 kg for site in South Korea) to 110 kg and body mass index (BMI) within the range 18 to 36 kg/m2, inclusive.
* For moderate hepatic impairment cohort: Child-Pugh total score ranging from 7 to 9, inclusive.
* For mild hepatic impairment cohort: Child-Pugh total score ranging from 5 to 6, inclusive

For matched subjects:

* Participant must be 40 to 75 years of age, inclusive.
* Female participants who are postmenopausal or are post-bilateral surgical oophorectomy not linked to a history of cancer. Menopause is defined as being amenorrheic for at least 12 months without an alternative medical cause, with plasma FSH level >30 IU/L or age ≥60 years.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Body weight within the range 50 kg (40 kg for site in South Korea) to 100 kg and body mass index (BMI) within the range 18 to 36 kg/m2, inclusive.

Exclusion Criteria:

For participants with hepatic impairment:

* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis) within 1 year before inclusion.
* Smoking regularly more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 8 cigarettes per day during the institutionalization (Smoking is not allowed within 8 hours after amcenestrant administration).
* Excessive consumption of beverages containing xanthine bases (more than 5 cups or glasses per day).
* Non-live vaccines including Covid-19: last administration of a vaccine within 1 week (symptoms-free) to 2 weeks before inclusion.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 72 hours before inclusion.
* Use of any herbal medicines 1 week before IMP administration and up to the end of PK sampling following the IMP administration
* Live-vaccines: last administration of a vaccine within 4 weeks before inclusion
* Treatment with a strong CYP3A, CYP2C8 or any UGTs inhibitor within 14 days before first study treatment administration or 5 half-lives whichever is longer.
* Treatment with a strong or moderate CYP3A, CYP2C8 or any UGTs inducer within 14 days before first study treatment administration or 5 half-lives whichever is longer.
* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic, renal, infectious disease, severe hepatic impairment (Child-Pugh total score greater than or equal to 10), or signs of acute illness, hepatocarcinoma, acute hepatitis, Hepatic encephalopathy Grade 2, 3, and 4
* Esophageal bleeding, which is caused by esophageal varices, within 3 months before inclusion

For matched subjects:

* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis) within 1 year before inclusion.
* Smoking regularly more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 8 cigarettes per day during the institutionalization (Smoking is not allowed within 8 hours after amcenestrant administration).
* Excessive consumption of beverages containing xanthine bases (more than 5 cups or glasses per day).
* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic, or infectious disease, or signs of acute illness, unless the Investigator considers an abnormality to be not clinically significant.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month.
* Non-live vaccines including Covid-19: last administration of a vaccine within 1 week (symptoms-free) to 2 weeks before inclusion
* Live-vaccines: last administration of a vaccine within 4 weeks before inclusion
* Treatment with a strong CYP3A, CYP2C8 or any UGTs inhibitor within 14 days before first study treatment administration or 5 half-lives whichever is longer.
* Treatment with a strong or moderate CYP3A, CYP2C8 or any UGTs inducer within 14 days before first study treatment administration or 5 half-lives whichever is longer.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 72 hours before inclusion.
* Use of any herbal medicines 1 week before IMP administration and up to the end of PK sampling following the IMP administration The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) assessment: Maximum plasma concentration observed (Cmax) | From Day 1 to Day 5
  Maximum plasma concentration observed (Cmax) of amcenestrant
PK assessment: Area under the plasma concentration (AUC) | From Day 1 to Day 5
  Area under the plasma concentration versus time curve of amcenestrant

SECONDARY OUTCOMES:
PK assessment: Tmax of amcenestrant | From Day 1 to Day 5
  Time to reach Cmax of amcenestrant
PK assessment: Area under the plasma concentration versus time curve (AUClast) of amcenestrant | From Day 1 to Day 5
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast of amcenestrant
PK assessment: Maximum unbound plasma concentration (Cmax u) of amcenestrant | From Day 1 to Day 5
  Maximum unbound plasma concentration of amcenestrant
PK assessment: AUCu of amcenestrant | From Day 1 to Day 5
  Unbound area under the plasma concentration versus time curve extrapolated to infinity of amcenestrant
PK assessment: Cmax of M7 | From Day 1 to Day 5
  Maximum observed plasma concentration of M7
PK assessment: AUClast of M7 | From Day 1 to Day 5
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast of M7
PK assessment: AUC of M7 | From Day 1 to Day 5
  Area under the plasma concentration versus time curve extrapolated to infinity of M7
Number of participants with adverse events (AEs) / treatment-emergent adverse events (TEAEs) | From the date when the ICF is signed to the end of study (approximately Day 10)
  Incidence of adverse events (AEs) and treatment-emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Investigational Site Number :2760001, Kiel, Germany
- South Korea (2):
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational site number :4100002, Cheongju-si

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: POP16301 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25331&tenant=MT_SNY_9011